CLINICAL TRIAL: NCT06118099
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Proof-of-concept Study Assessing the Efficacy and Safety of Amlitelimab in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Proof-of-concept Study Evaluating Subcutaneous Amlitelimab in Adult Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision; the decision is not related to any safety concern
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17967; U1111-1290-9497 (Registry Identifier: ICTRP); 2023-505803-22 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis
MeSH Terms: conditions — Hidradenitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Amlitelimab (Experimental): Subcutaneous injection (SC) as per protocol.
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Injection solution SC injection
  Other Names: SAR445229
  Arms: Amlitelimab
Drug: Placebo — Injection solution SC injection
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2, 2-arm, double-blind, randomized, multicenter, multinational, placebo-controlled study to evaluate efficacy, safety, pharmacokinetics (PK), and biological effects of treatment of subcutaneous injection of amlitelimab compared with placebo in male and female participants aged 18 to 70 years with moderate to severe hidradenitis suppurativa (HS).

The purpose of this study is to measure standardized clinician reported and participant-reported outcomes (ClinRO and PRO), safety, and drug concentration. An optional long-term extension (LTE) period will assess chronic safety and efficacy over an additional 80 weeks of amlitelimab treatment.

Study details include:

* The study duration will be up to 116 weeks, including a 4-week Screening period, a 16-week double-blind treatment period (DBT), an optional 80-week LTE period and a 16-week post-treatment follow-up period.
* All participants who complete the 16-week DBT period will be offered entry into an optional LTE.
* Participants who do not wish to enter the optional LTE period or who stop treatment prior to Week 16 (Visit 6) or stop investigational medicinal product (IMP) administration prior to completing the LTE period will proceed into the 16-week post-treatment follow-up period.
* The number of planned in clinic visits will be up to six during the DBT period with an additional nine during the LTE period, plus one post-treatment follow-up end-of-study visit. Up to 11 optional in clinic visits are allowed for participants who do not wish to self-administer IMP between scheduled in clinic visits during the LTE period.

DETAILED DESCRIPTION:
The study duration per participant will be up to 116 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 (or country's age of majority if >18) years to 70 years of age inclusive, at the time of signing the informed consent.
* Participants with a history of signs and symptoms consistent with HS for at least 1 year prior to baseline.
* Participants must have HS lesions present in at least 2 distinct anatomic areas (eg, left, and right axilla; or left axilla and left inguino-crural fold), 1 of which must be Hurley Stage II or Hurley Stage III.
* Participant must have had an inadequate response to at least a 12-week trial of an oral antibiotic for treatment of HS

Exclusion Criteria:

* Participants with a diagnosis of inflammatory conditions other than HS (including but not limited to systemic lupus erythematosus, systemic sclerosis, myositis, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, multiple sclerosis, Behcet's disease, sarcoidosis, etc)
* Any other active skin disease or condition (eg, bacterial, fungal, or viral infection) that may interfere with assessment of HS

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
The clinical response as measured by the percentage of participants achieving HiSCR50 at Week 16 | Week 16
  Hidradenitis suppurativa clinical response (HiSCR)50 is defined as ≥50% reduction from baseline in the total abscess and inflammatory nodule count (AN count), with no increase from baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Time to onset of achieving HiSCR50 | From baseline to Week 16
  HiSCR50 is defined as ≥50% reduction from baseline in the total abscess and inflammatory nodule count (AN count), with no increase from baseline in abscess or draining tunnel count.
Absolute change from baseline in AN count at Week 16 | Baseline to Week 16
  AN count is the total abscess and inflammatory nodule count.
Percentage change in AN count at Week 16 | Baseline to Week 16
  AN count is the total abscess and inflammatory nodule count.
Percentage of participants achieving HiSCR75 at Week 16 | Week 16
  HiSCR75 is defined as ≥75% reduction from baseline in the total abscess and inflammatory nodule count (AN count), with no increase from baseline in abscess or draining tunnel count.
Percentage of participants achieving HiSCR90 at Week 16 | Week 16
  HiSCR90 is defined as ≥90% reduction from baseline in the total abscess and inflammatory nodule count (AN count), with no increase from baseline in abscess or draining tunnel count.
Percentage of participants who experience improvement by at least 1 International Hidradenitis Suppurativa Severity Score System (IHS4) stage at Week 16 | Week 16
  The IHS4 is a validated tool to assess HS severity. A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.
Change in absolute score from Baseline in IHS4 at Week 16 | Baseline to Week 16
  The IHS4 is a validated tool to assess HS severity. A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.
Percentage of participants who experience a flare at Week 16 | Week 16
  A flare is defined as at least a 25% increase in AN count (with a minimum increase of 2 AN) relative to baseline. AN count is the total abscess and inflammatory nodule count.
Percentage of participants achieving IHS4-55 at Week 16 | Week 16
  IHS4-55 is defined as achievement of a 55% reduction in IHS4 score from baseline. A total score of 3 or less signifies mild, 4 to 10 signifies moderate, and 11 or higher signifies severe disease.
Percentage of participants achieving at least 30% reduction and at least 1 unit reduction from Baseline in weekly average of daily HS-Skin Pain NRS at Week 16 among participants with baseline NRS ≥3 | Week 16
  Hidradenitis Suppurativa-Skin pain-numeric rating scale (HS-Skin pain NRS) is scored on a 0 to 10 scale with 0 indicating "no skin pain" and 10 indicating "worst skin pain possible".
Percentage of participants with improvement (reduction) in Peak Pruritus Numerical Rating Scale (PP-NRS) ≥4 from Baseline at Week 16 among participants with baseline PP-NRS ≥4 | Week 16
  PP-NRS is a validated single item 0 (no itch) to10 (worst itch imaginable) numeric rating scale assessing peak pruritus (itch).
Percentage of participants who experience 5-point reduction in DLQI at Week 16 among participants with baseline DLQI ≥4 | Week 16
  Dermatology life quality index (DLQI) is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL). Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Change from Baseline in the total Hidradenitis Suppurativa Quality of Life (HiSQOL) score at Week 16 | Baseline to Week 16
  HiSQOL is an instrument designed to measure the HS-specific health-related QoL of adults with HS.
Incidence of treatment-emergent adverse events (TEAEs), adverse event of special interest (AESIs), and serious adverse events (SAEs) including local injection site reactions in the Safety Population | Baseline up to Week 116
Incidence of potentially clinically significant abnormalities in laboratory tests, vital signs, and electrocardiograms in the Safety Population | Baseline up to Week 116
Serum amlitelimab concentrations measured at prespecified time points in the PK population | Day 1 up to Week 116
Incidence of antidrug antibodies (ADA) of amlitelimab at prespecified timepoints in the ADA population | Day 1 up to Week 116

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (42):
- United States (12):
  - Medical Dermatology Specialists Site Number : 8400002, Phoenix, Arizona
  - Center for Dermatology Clinical Research Site Number : 8400010, Fremont, California
  - Corazon USA, LLC (DBA Life Clinical Trials) Site Number : 8400011, Margate, Florida
  - Florida International Research Center Site Number : 8400016, Miami, Florida
  - University of South Florida Site Number : 8400012, Tampa, Florida
  - Beth Israel Deaconess Medical Center Site Number : 8400006, Boston, Massachusetts
  - Washington University School of Medicine Site Number : 8400007, St Louis, Missouri
  - Centricity Research Site Number : 8400009, Dublin, Ohio
  - Clinical Partners, LLC Site Number : 8400003, Johnston, Rhode Island
  - Vast Skin Specialists Site Number : 8400015, Addison, Texas
  - Center for Clinical Studies, LTD. LLP Site Number : 8400001, Houston, Texas
  - Stryde Research Epiphany Dermatology Site Number : 8400014, Southlake, Texas
- Australia (3):
  - Investigational Site Number : 0360003, Phillip, Australian Capital Territory
  - Investigational Site Number : 0360001, Darlinghurst, New South Wales
  - Investigational Site Number : 0360002, Melbourne, Victoria
- Canada (3):
  - Investigational Site Number : 1240007, Barrie, Ontario
  - Investigational Site Number : 1240002, Hamilton, Ontario
  - Investigational Site Number : 1240001, Québec
- Chile (3):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- France (5):
  - Investigational Site Number : 2500005, La Rochelle
  - Investigational Site Number : 2500003, Lyon
  - Investigational Site Number : 2500001, Reims
  - Investigational Site Number : 2500004, Rouen
  - Investigational Site Number : 2500002, Saint-Mandé
- Germany (2):
  - Investigational Site Number : 2760002, Bochum
  - Investigational Site Number : 2760001, Münster
- Hungary (3):
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480001, Debrecen
  - Investigational Site Number : 3480002, Szeged
- Italy (2):
  - Investigational Site Number : 3800001, Catania
  - Investigational Site Number : 3800002, Cona (Ferrara)
- Poland (3):
  - Investigational Site Number : 6160001, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160004, Warsaw
  - Investigational Site Number : 6160003, Wroclaw
- Portugal (2):
  - Investigational Site Number : 6200002, Lisbon
  - Investigational Site Number : 6200001, Lisbon
- Spain (4):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240006, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17967 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25516&tenant=MT_SNY_9011